CLINICAL TRIAL: NCT07248332
Title: The Efface of Lidocaine vs. Magnesium Sulphate in the Management of Pain After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Efface of Lidocaine vs. Magnesium Sulphate in the Management of Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Mustafa Hussain Imam, Mustafa Hussain Imam, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1095-2024-LNH-ERC
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Cholecystectomy Surgery; Postoperative Pain Management
Keywords: Lidocaine; Magnesium Sulphate; Postoperative Pain; Laparoscopic Cholecystectomy; Visual Analogue Scale (VAS); analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulphate Group (Active Comparator): The magnesium sulfate dose was prepared as 2 mg, diluted with normal saline to a total volume of 10 mL, and administered intravenously as a single stat dose at the time of anesthesia reversal after completion of surgery.
  Interventions: Drug: IV 2mg of Magnesium Sulphate
- Lidocaine Group (Active Comparator): A total of 3 mL of 2% lidocaine was combined with 7 mL of normal saline to prepare a 10 mL solution, which was given intravenously as a single stat dose at the time of anesthesia reversal immediately after the surgery was completed.
  Interventions: Drug: IV Lidocain 60 mg/kg

INTERVENTIONS:
Drug: IV 2mg of Magnesium Sulphate — Patients in the magnesium sulfate group received 2 mg of the drug, which was diluted with normal saline to a total volume of 10 mL and administered intravenously as a single stat dose at the time of anesthesia reversal following completion of laparoscopic cholecystectomy. The injection was performed under aseptic conditions by an anesthetist who was blinded to group assignment. All participants received routine postoperative care, including intravenous diclofenac sodium 75 mg every 8 hours for baseline pain control and intravenous ondansetron 4 mg to prevent nausea. Postoperative pain intensity was measured using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours. Patients experiencing significant pain were given intravenous Kinz 5 mg as rescue analgesia, and the timing of administration was recorded for documentation.
  Arms: Magnesium Sulphate Group
Drug: IV Lidocain 60 mg/kg — Patients in the Lidocaine group received 3 mL of 2% lidocaine, diluted with 7 mL of normal saline to prepare a 10 mL solution, which was administered intravenously as a stat dose at the time of anesthesia reversal, immediately after surgery. The intervention was given using the same protocol and blinding method as the Ketamine group to maintain uniformity. Similar to Group K, all patients received standard postoperative medications, including IV diclofenac sodium and ondansetron. Pain assessment was performed using the VAS scale at 1, 6, 12, and 24 hours postoperatively. Patients requiring additional pain relief were given IV Kinz 5 mg as rescue analgesia, with the time of each administration noted.
  Arms: Lidocaine Group

SUMMARY:
This prospective interventional study was carried out at Liaquat National Hospital and Medical College to evaluate and compare the postoperative analgesic effects of intravenous lidocaine and magnesium sulphate in patients undergoing laparoscopic cholecystectomy. A total of 168 ASA I-II patients were enrolled and randomly allocated into two groups of 84 participants each (Group L: Lidocaine, Group M: Magnesium Sulphate) using a sealed-envelope randomization technique in a double-blind, placebo-controlled design. All patients received standardized general anesthesia with propofol, isoflurane, and atracurium, and routine postoperative care included intravenous diclofenac sodium and ondansetron. Postoperative pain was measured at 1, 6, 12, and 24 hours using the Visual Analogue Scale (VAS) to assess and compare the efficacy and duration of analgesia between the two groups. The study aimed to provide insight into the relative analgesic performance of lidocaine and magnesium sulphate, supporting improved pain management strategies following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Optimal management of postoperative pain is crucial for enhancing recovery, minimizing stress responses, and promoting better outcomes after laparoscopic cholecystectomy. This prospective interventional study was carried out in the Department of Anesthesiology at Liaquat National Hospital and Medical College to compare the analgesic effects of intravenous lidocaine and magnesium sulphate in patients undergoing elective laparoscopic cholecystectomy.

A total of 168 patients classified as ASA I-II with uncomplicated symptomatic gallstones were enrolled after obtaining ethical approval and written informed consent. Participants were randomly assigned into two equal groups of 84 patients each (Group L: Lidocaine, Group M: Magnesium Sulphate) using a sealed-envelope technique. The study employed a double-blind, placebo-controlled design to ensure unbiased evaluation. Patients with ASA III-V, chronic pain disorders, psychiatric conditions, pregnancy or breastfeeding, major hepatic, renal, or cardiovascular disease, or recent use of opioids or NSAIDs were excluded from the study.

All patients underwent standard preoperative assessment, including overnight fasting and anesthetic evaluation. General anesthesia was induced with propofol and atracurium and maintained with isoflurane. Intraoperative monitoring included heart rate, blood pressure, ECG, oxygen saturation, and end-tidal CO₂. Residual neuromuscular blockade was reversed with neostigmine at the end of surgery. Postoperative care included intravenous diclofenac sodium every 8 hours for baseline analgesia and ondansetron for prevention of nausea and vomiting.

Postoperative pain intensity was recorded at 1, 6, 12, and 24 hours using the Visual Analogue Scale (VAS). Patients experiencing significant pain were administered intravenous Kinz 5 mg as rescue analgesia, and the timing was documented by nursing staff.

This study provided important information on the comparative efficacy of lidocaine and magnesium sulphate for postoperative pain management, highlighting their potential role in multimodal analgesic strategies to improve patient comfort and recovery following laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years. ASA physical status I-II. Elective laparoscopic cholecystectomy planned under general anesthesia. Normal baseline renal, hepatic, and coagulation profile. Able to give informed consent and communicate pain scores. Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* • ASA III-V patients. Allergy or hypersensitivity to ketamine, lidocaine, or related drugs. History of psychiatric illness or substance abuse. Chronic use of opioids, benzodiazepines, or MAO inhibitors. Pregnant or breastfeeding women. Chronic pain disorders or use of analgesics within 7 days pre-op. Major hepatic, renal, or cardiovascular dysfunction. History of myopathy or seizure disorders. Patients with atrioventricular block or on calcium-channel blockers. Conversion to open cholecystectomy during surgery. Inability to understand or report pain postoperatively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Postoperative pain was assessed at the 1st, 6th, 12th, and 24th hours.
  Postoperative pain intensity was assessed using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours after surgery to evaluate and compare the effectiveness and duration of analgesia between the ketamine and lidocaine groups. These time intervals were selected to monitor both the early and late postoperative pain responses during the first 24 hours of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Hussain Imam, MBBS, Principal Investigator — Liaquat National Hospital; Ali Asgher, Mbbs, FCPS, Study Director — Liaquat National Hospital
Locations (1):
- Anesthesiology Department Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No